CLINICAL TRIAL: NCT03852303
Title: OAETREAT Extra Ivermectin Treatment of Persons With Onchocerciasis-associated Epilepsy: a
Brief Title: Ivermectin Treatment of Persons With Onchocerciasis-associated Epilepsy
Acronym: OAETREATe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Robert Colebunders, Prof, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B300201733349
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ivermectin once a year (Active Comparator): Ivermectin one dose per year and anti-epileptic treatment
  Interventions: Drug: ivermectin
- ivermectin 2 times a year (Experimental): Ivermectin one dose 2 times a year and anti-epileptic treatment
  Interventions: Drug: ivermectin
- ivermectin 3 times a year (Experimental): vermectin one dose 3 times a year and anti-epileptic treatment
  Interventions: Drug: ivermectin

INTERVENTIONS:
Drug: ivermectin — evaluate effect of ivermectin on frequency of seizures
  Other Names: anti-epileptic treatment

SUMMARY:
Randomized clinical trial in the Logo health zone, in Ituri province, Democratic Republic of Congo to compare seizure freedom in onchocerciasis infested epilepsy patients who ivermectin treatment once a year compared to 2 and 3 times a year. All participants also receive anti-epileptic drugs according to local guidelines for epilepsy treatment. Participants will be followed for 12 months. The primary endpoint is seizure freedom defined as no seizures during the last fourth months of the trial.

DETAILED DESCRIPTION:
Randomized clinical trial in the Logo health zone, in Ituri province, Democratic Republic of Congo to compare seizure freedom in onchocerciasis infested epilepsy patients who ivermectin treatment once a year compared to 2 and 3 times a year. All participants also receive anti-epileptic drugs according to local guidelines for epilepsy treatment. Participants will be followed for 12 months.The primary endpoint is seizure freedom defined as no seizures during the last fourth months of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years and above
* Signed informed consent form
* Normal neurological development until onset of epilepsy
* Onset of epilepsy between ages of 5 and 18 years
* Presence of microfilaria in skin snip and/or antibodies against Ov16

Exclusion Criteria:

* Ivermectin intake the last 9 months
* Pregnancy or breastfeeding
* Known or suspected allergy to Ivermectin
* Loa Loa microfilariae in blood
* Epilepsy with known cause (e.g. severe head trauma, perinatal asphyxia, patients with a history of cerebral malaria, meningitis or encephalitis)
* Concomitant acute illness or chronic medication use
* Chronic alcohol/substance use

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
seizure freedom | month 9-12
  no seizures

CONTACTS AND LOCATIONS:
Overall Officials: Robert Colebunders, MD,PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Centre de Recherche en Maladies Tropicales de l'Ituri, Rethy, Ituri, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
A
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of results
Access Criteria: Approval of the PI